CLINICAL TRIAL: NCT02153242
Title: Does a Surrogate Marker Exist That Can be Used as A Predictor For Left Ventricular Dysfunction In Patients Undergoing Right Ventricular Pacing
Brief Title: The Effects of Selective Site Right Ventricular Pacing
Acronym: PacingRV
Status: Completed | Type: Observational
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: B596
Record Dates: First submitted 2014-05-06; First posted 2014-06-03 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Bradycardia
Keywords: Pacing; Haemodynamics; Pilot
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Supra Ventricular Tachycardia (SVT): Patients undergoing SVT studies

SUMMARY:
This is a pilot study into the effects on heart function when pacing the right ventricle (RV). This study aims to enrol a population with structurally normal hearts. The investigators aim to measure heart function directly when pacing.

When normal conduction within the heart fails, the treatment may be to implant a permanent pacemaker. Pacing involves passing a lead via a vein to the heart and using an electrical impulse to stimulate a beat. The usual site for pacing is the tip of the RV. This has been shown to be less efficient than the normal conduction system of the heart and in some cases leads to markedly reduced function. What the investigators do not know is why this is the case.

Much effort has been directed at looking at features within the left ventricle (LV) for markers of disease progression but little has been investigated regarding the RV.

There may be some benefit to pacing the heart preferentially from different parts of the RV and the investigators aim to measure if any differences are detectable from stimulating the heart at various sites within the RV.

DETAILED DESCRIPTION:
Inclusion Criteria;

* Patients undergoing elective Electrophysiological Studies +/Ablation
* Age 18-80
* Normal Heart on Pre-procedural Echocardiogram

Exclusion criteria;

* Atrial Fibrillation
* Evidence of anterograde conducting accessory pathway
* Permanent Pacemaker insitu
* Pregnant
* Breast Feeding

Outcome Measures; Change in load-independent indices of LV and RV contractility before and after pacing intervention. LV and RV function measured by transthoracic echocardiography and tissue Doppler imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective Electrophysiological Studies +/Ablation
* Age 18-80
* Normal Heart on Pre-procedural Echocardiogram

Exclusion criteria:

* Atrial Fibrillation
* Evidence of anterograde conducting accessory pathway
* Permanent Pacemaker insitu
* Pregnant
* Breast Feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing SVT studies
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Ventricular Function | 30 minutes
  Measurement of both right and left ventricular function under differing pacing conditions

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Tan, Principal Investigator — Basildon & Thurrock University Hospital NHS Trust
Locations (1):
- The Essex Cardiothoracic Centre, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No